CLINICAL TRIAL: NCT02726516
Title: Effects of PRJ-205 on Performance in Trained Young Subjects After Acute and Chronic Intake of the Study Product
Brief Title: Effects of PRJ-205 on Performance in Trained Young Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioiberica (Industry)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: PRJ-205
Record Dates: First submitted 2016-03-23; First posted 2016-04-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated (Experimental): Treated volunteers will be administered one dose of PRJ-205 1,5 hours before the exercise task for the acute testing and will be taking one dose per day of PRJ-205 for 4 days for the chronic testing.
  Interventions: Dietary Supplement: PRJ-205
- Placebo (Placebo Comparator): Placebo volunteers will be administered one dose of placebo 1,5 hours before the exercise task for the acute testing and will be taking one dose per day of placebo for 4 days for the chronic testing.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: PRJ-205 — 1 sachet per day
  Arms: Treated
Other: Placebo — 1 sachet per day
  Arms: Placebo

SUMMARY:
Compare a dietary supplement (PRJ-205) and placebo during 1 or 4 days on aerobic exercise performance, oxidative stress and muscle damage.

The hypothesis is that supplementation with PRJ-205 improve aerobic performance

DETAILED DESCRIPTION:
Twenty young active males will be recruited and randomized to either placebo or PRJ-205. Subjects will take the designated treatment in an acute dosage and chronically, 4 days of treatment.

They will undergo 3 exercise tasks (before the administration of the product, 1.5h after the acute administration of the product and after 4 days of treatment). VO2max and anaerobic threshold will be measured during the tests. Blood samples will be taken to measure muscle damage and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Physically active

Exclusion Criteria:

* known cardiovascular, pulmonary or metabolic disease
* any medical condition that could affect the development and safety of the exercise task

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Aerobic performance determined by VO2max | 4 days

SECONDARY OUTCOMES:
Pressure pain threshold of calf muscle | 4 days
  Measured pre- and post- exercise task
Serum markers of muscular damage | 4 days
  Measured from blood samples taken pre- and post- exercise task.
Oxidative stress parameters | 4 days
  Measured from blood samples taken pre- and post- exercise task.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Viña, PhD, Principal Investigator — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided